CLINICAL TRIAL: NCT04654481
Title: Feasibility of Using a Home-Based High Frequency Chest Wall Oscillation Device (AffloVest) in At-Risk Respiratory Patients to Decrease Acute Respiratory Care Burden During the COVID-19 Pandemic
Brief Title: Study of AffloVest in At-Risk Respiratory Patients During COVID-19 Pandemic
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: only one participant enrolled, results will not be provided due to risk of breach of confidentiality
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: International Biophysics Corporation (Industry); SPARK Healthcare (Unknown)
Responsible Party: Principal Investigator, Patricia Walker, Co-Director, The Cystic Fibrosis Center, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 20-2667; ISMMS-AFF-20 (Other: International Biophysics, Inc.)
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Cough; Covid19
Keywords: Pulmonary Disease; Airway Clearance Therapy; High Frequency Chest Wall Oscillation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Chronic Cough; COVID-19; Lung Diseases | interventions — Chest Wall Oscillation; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician and data analysts will be blinded to treatment cohort.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Care Plus Monitoring (Active Comparator): All subjects will be monitored via home spirometry, pulse oximetry, temperature checks, telehealth check-in and patient-reported outcome assessments.
  Interventions: Other: Standard Care Plus Monitoring
- Standard Care Plus Monitoring and HCFWO (Experimental): In addition to home spirometry, pulse oximetry, temperature checks, telehealth check-in and patient-reported outcome assessments, subject will receive an Afflovest device for home use.
  Interventions: Device: HCFWO; Other: Standard Care Plus Monitoring

INTERVENTIONS:
Device: HCFWO — The Afflovest device is a High Frequency Chest Wall Oscillation (HFCWO) device, a medical vest that uses vibrations to loosen and mobilize mucus in the lung secretions and help clear the airways.
  Other Names: High Frequency Chest Wall Oscillation; Afflovest
  Arms: Standard Care Plus Monitoring and HCFWO
Other: Standard Care Plus Monitoring — Monitoring via home spirometry, pulse oximetry, temperature checks, telehealth check-in and patient-reported outcome assessments.

SUMMARY:
The purpose of the study is to investigate the addition of high frequency chest wall oscillation (HFCWO) therapy to the prescribed care regimen to support the diaphragm during airway clearance among post-COVID patients with COPD and chronic productive cough as a way to limit the advancement of pulmonary symptoms and need for critical services during recovery from COVID-19.

DETAILED DESCRIPTION:
Thirty study participants in New York City who meet inclusion criteria will be recruited from Mount Sinai's COVID-19 Post-Recovery Center of Excellence and Respiratory Institute. Fifteen subjects (determined by the last digit of their medical record number) will receive a HFCWO device (AffloVest), digital thermometer, pulse oximeter, and spirometer at their home. Participants will be trained remotely to use the AffloVest and spirometer. In addition all subjects will be asked to complete a series of online mental health and respiratory symptom assessments via REDCap. A 15 patient control group meeting inclusion criteria will be recruited from the Mount Sinai COVID-19 Post-Recovery Center of Excellence and Respiratory Institute using the same screening process. This group will not receive the HFCWO intervention but will receive a digital thermometer, pulse oximeter, and spirometer at their home (with training via telehealth), asked to complete all REDCap and respiratory symptom assessments. Consent for both groups will be obtained by a Mount Sinai clinician-researcher.

Study Duration Approximately 30 days plus 60 and 90-day check in

Objectives To investigate the addition of HFCWO therapy to the prescribed care regimen to support the diaphragm during airway clearance among post-COVID patients with COPD and chronic productive cough as a way to limit the advancement of pulmonary symptoms and need for critical services during recovery from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females ≥18 years
* Existing diagnosis of COPD for >6 months
* Chronic productive cough
* Radiographic evidence of flattening of the diaphragm
* Prior COVID-19 diagnosis
* Clinically followed by Mount Sinai COVID-19 Post Recovery and Respiratory Institute.
* Ability to provide informed consent
* Ability to read and fill out survey questionnaires via REDCap (surveys will be available in English and Spanish)
* Access to a home computer, tablet, or smartphone

Exclusion Criteria:

* Presenting with hypoxia (02 sat <90%)
* Acute COVID-19 infection
* Home oxygen dependent
* Established diagnosis of cystic fibrosis
* History of osteoporosis or rib fracture
* Active Hemoptysis
* Pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in one second (FEV1) | Baseline and up to 90 Days
  Change in forced expiratory volume in one second (FEV1) as compared to baseline, measured by home spirometer.
Change in Oxygen Saturation level | Baseline and up to 90 Days
  Changes in oxygen saturation from baseline as measured by pulse oximeter. Normal oxygen range is 95 to 100 percent and low oxygen range is under 90 percent.
Change in Presence of Fever | Baseline and up to 90 Days
  Changes in basal temperature as measured by digital thermometer. Fever is indicated at 100.4 F (38 C) or higher.

SECONDARY OUTCOMES:
Change in Presence of pneumonia symptoms via Community Acquired Pneumonia (CAP) Symptom Questionnaire | Baseline and up to 90 Days
  CAP Symptom Questionnaire records how much the patient rated the bothersomeness of the symptom. Each item is scored as "0" (Patient did not have this symptom), "1" (Not at All) to "5" (Extremely). Full range scale from 0 to 90, higher score indicating patient experiencing more frequent or more severe symptoms.
Change in Quality of life via Quality of Life Questionnaire-Respiratory (QOL-B) | Baseline and up to 90 Days
  The QOL-B is a disease-specific questionnaire that measures symptoms, functioning, and health-related quality of life relevant to patients with bronchiectasis. Scores are generated from 37 items that fall on 8 domains: Physical Functioning, Role Functioning, Vitality, Emotional Functioning, Social Functioning, Treatment Burden, Health Perceptions, and Respiratory Symptoms. All subscales and the full range scale are standardized to score from 0 to 100, with higher scores indicating better enjoyment and satisfaction with specific life domains.
Change in Mental health screening via Personal Health Questionnaire Depression Scale (PHQ-8) | Baseline and up to 90 Days
  The PHQ-8 is the depression module, which scores each of the eight DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Full scale from 0-24, with higher score indicating more severe symptoms.
Change in Mental health screening via General Anxiety Disorder-7 (GAD-7) | Baseline and up to 90 Days
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). Full scale from 0-21, with higher score indicating more symptoms.
Change in COVID Symptom Checklist | Baseline and up to 90 Days
  Eight questions that are specific to recent literature describing patients' experiences of symptoms during COVID. They are rated on a frequency scale from "never" to "always," using a 1-4 point scale. Full scale range from 8 to 32, with higher scores indicating more frequent symptoms.
AffloVest Usage | 90 Days
  Amount of time used per week in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Beth Israel, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No